CLINICAL TRIAL: NCT06995625
Title: An Open-Label, Single-Arm, Dose Escalation Phase I Clinical Trial to Evaluate the Safety and Tolerability of SNE-101 in Patients With Acute Ischemic Stroke
Brief Title: The STem Cell-derived Extracellular Vesicle Therapy In Acute Ischemic Stroke (STEVIA)
Acronym: STEVIA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: S&Ebio Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNE-101S
Record Dates: First submitted 2025-05-13; First posted 2025-05-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke AIS
Keywords: Stroke; Exosome; Extracellular vesicles; Wharton's jelly-mesenchymal stem cell; MSC
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SNE-101 (Experimental): Patients will be given SNE-101, an extracellular vesicle derived from Wharton's jelly mesenchymal stem cells.
  • Drug: SNE-101
  * Three multiple doses of SNE-101 will be administered to three study cohorts , each consisting of 3 to 6 subjects.
  * SNE-101 will be administered intravenously once a day for 5 days.
  Interventions: Drug: SNE-101

INTERVENTIONS:
Drug: SNE-101 — Experimental: Cohort 1 - SNE-101 4.8 × 10e10 particles (n=3 to 6) Experimental: Cohort 2 - SNE-101 9.6 × 10e10 particles (n=3 to 6) Experimental: Cohort 3 - SNE-101 19.2 × 10e10 particles (n=3 to 6)

SUMMARY:
This is a multicenter open-label, single-arm, dose escalation phase I clinical trial to evaluate the safety and tolerability of SNE-101 in patients with acute ischemic stroke

DETAILED DESCRIPTION:
The study aims to assess the safety, tolerability, and preliminary efficacy of allogeneic Wharton's jelly-mesenchymal stem cell-derived extracellular vesicles (EVs) in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults with 19 years or older
* Patients within 5 days of symptom onset who have not received thrombolytic therapy or undergone endovascular reperfusion procedures.
* Patients within 5 days of symptom onset who have received thrombolytic therapy or undergone endovascular reperfusion procedures but show no clinical recovery after 2 days of observation.
* Imaging findings must meet both of the following:

  * Infarction within the middle cerebral artery territory on diffusion-weighted imaging (DWI)
  * Infarct size ≥ 20 mm in the longest diameter on DWI
* Neurological status meeting all three of the following NIHSS criteria:

  * Moderate to severe neurological deficit (NIHSS score between 5-21)
  * New onset of motor weakness (score 2-4 in at least one of NIHSS items 5a, 5b, 6a, or 6b)
  * No impaired consciousness (score 0-1 on NIHSS items 1a, 1b, and 1c)
* Voluntary written informed consent

Exclusion Criteria:

Subjects are ineligible if they meet any of the following:

* Pre-stroke disability (pre-stroke mRS ≥ 2)
* Likely to recover spontaneously, based on all three of:

  * No longer meeting the NIHSS inclusion criteria 48 hours post-thrombolysis or endovascular therapy
  * Lacunar stroke due to small vessel occlusion
  * SAFE (Shoulder Abduction and Finger Extension) score ≥ 5
* Presence or risk of malignant middle cerebral artery infarction with brain edema
* Significant medical history within the past 5 years:

  * Severe heart failure
  * Severe infectious disease
  * Severe hepatic failure or renal failure
  * Newly diagnosed or actively treated cancer
  * Any systemic disease deemed by investigator to significantly reduce life expectancy
  * Any condition likely to hinder follow-up during the study
* Diagnosed severe psychiatric illness:

  * Moderate or greater depression pre-stroke with functional impairment and suicide risk
  * Pre-stroke dementia interfering with daily living (CDR ≥ 2)
* Contraindication to MRI (e.g., pacemaker)
* Pregnant or breastfeeding, or unwilling to use effective contraception method for 90 days after last dose.
* Participation in another clinical trial within the past 3 months
* Any other reason determined by the investigator that would prevent participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SNE-101 in patients with acute ischemic stroke and determine the Maximum Tolerated Dose (MTD) | MTD: within 19 days after first dose
  o The Maximum Tolerated Dose (MTD) determination via the Dose limiting toxicity (DLT)
To evaluate the safety and tolerability of SNE-101 in patients with acute ischemic stroke and determine the Maximum Tolerated Dose (MTD) | Adverse events: 180 days
  o Adverse events are monitored continuously throughout the study.

SECONDARY OUTCOMES:
To assess the efficacy of SNE-101 in patients with acute ischemic stroke. | 13 weeks
  o Mean % change in Fugl-Meyer Assessment (FMA) from baseline to Week 13
  A quantitative measure used to assess motor function, balance, and joint motion in post-stroke patients. The FMA is a widely validated scale used to evaluate sensorimotor recovery, especially in the upper and lower extremities, with a maximum score of 226 indicating normal function. Higher scores indicate better motor recovery.
To assess the efficacy of SNE-101 in patients with acute ischemic stroke. | 13 weeks
  o Improvement in neural tract integrity on Diffusion Tensor Imaging (DTI) from baseline to Week 13.
  An advanced MRI technique used to assess the integrity and organization of white matter tracts in the brain. DTI parameters such as fractional anisotropy (FA) and mean diffusivity (MD) provide quantitative measures of axonal regeneration and neuroplasticity. Increases in FA and normalization of MD values are indicative of neural recovery after stroke.
To assess the efficacy of SNE-101 in patients with acute ischemic stroke. | 13 weeks
  o Changes in NIH stroke scale (NIHSS) from baseline to Week 13
  A standardized neurological examination that quantifies the severity of neurological impairment caused by stroke. The NIHSS evaluates several domains including consciousness, motor strength, language, vision, and sensory loss. Scores range from 0 to 42, with lower scores indicating milder neurological deficits.
To assess the efficacy of SNE-101 in patients with acute ischemic stroke. | 13 weeks
  o Changes in modified Rankin Score (mRS) from baseline to Week 13
  A global functional outcome scale that assesses the degree of disability or dependence in daily activities in patients who have suffered a stroke. Scores range from 0 (no symptoms) to 6 (death). Lower scores indicate greater functional independence and are commonly used as primary endpoints in stroke trials.
To assess the efficacy of SNE-101 in patients with acute ischemic stroke. | 13 weeks
  o Changes in Infarct size from baseline to Week 13
  The volume of cerebral infarction measured using MRI sequences such as diffusion-weighted imaging (DWI) and fluid-attenuated inversion recovery (FLAIR). Reduction in infarct growth or final infarct size is considered an imaging biomarker of neuroprotection. Measurements are expressed in cubic centimeters (cc) and compared over time to assess treatment efficacy.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Ewha Womans University Seoul Hospital, Seoul